CLINICAL TRIAL: NCT01449344
Title: Efficacy and Safety of Rituximab, High-dose Ara-C and Dexamethasone (R-HAD) Alone or in Combination With Bortezomib in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Efficacy and Safety of R-HAD Alone or in Combination With Bortezomib in Patients With Relapsed or Refractory MCL
Acronym: (R-HAD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. M. Dreyling (co-chairman) (Other)
Collaborators: Klinikum der Universitaet Muenchen, Grosshadern (Other); ClinAssess GmbH (Industry); GELARC Service de Pharmacovigilance, Pierre Benite (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. M. Dreyling (co-chairman), Coordinating investigator, Germany, European Mantle Cell Lymphoma Network
Organization: European Mantle Cell Lymphoma Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCL2005-01
Record Dates: First submitted 2011-09-28; First posted 2011-10-10 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Mantle Cell Lymphoma
Keywords: relapsed; refractory
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — Rituximab; Cytarabine; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- R-HAD + Bortezomib (Experimental)
  Interventions: Drug: Rituximab; Drug: High dose Ara-C; Drug: Dexamethasone; Drug: Bortezomib
- R-HAD (Active Comparator)
  Interventions: Drug: Rituximab; Drug: High dose Ara-C; Drug: Dexamethasone

INTERVENTIONS:
Drug: Rituximab — Rituximab 375mg/m² IV , day 1
  Other Names: Rituximab:Rituxan
Drug: High dose Ara-C — Ara-C 2000 mg/m² (patients >65 years or s/p myeloablative treatment: 1000 mg/m²) IV, d 2 and 3
  Other Names: Ara-C: Cytarabine
Drug: Dexamethasone — Dexamethasone 40 mg PO, day 1-4
  Other Names: Dexamethasone: none
Drug: Bortezomib — Bortezomib 1.5 mg/m² IV, day 1 and 4
  Other Names: Bortezomib: Velcade
  Arms: R-HAD + Bortezomib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of rituximab, high-dose ara-c and dexamethasone (r-had) alone or in combination with bortezomib in patients with relapsed or refractory mantle cell lymphoma.

DETAILED DESCRIPTION:
This study is a prospective, randomized, multicenter, open-label phase III clinical trial to compare the efficacy and safety of Bortezomib in combination with Rituximab, high-dose Ara-C and dexamethasone (R-HAD) to R-HAD alone in patients with relapsed or refractory MCL after or not eligible for myeloablative treatment. The primary endpoint is time to treatment failure (TTF). Secondary endpoints are the complete response (CR) rate, the overall response (CR,PR) rate, the progression-free survival (PFS), the progression free survival of responders, the time to next lymphoma treatment, overall survival (OS), safety and tolerability of Rituximab, high-dose Ara-C and dexamethasone alone or in combination with Bortezomib. Study arms will be compared to each other to evaluate the impact of additional Bortezomib. Study arms will also be compared to historical controls.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathological diagnosis of MCL according to WHO classification.
* Relapse or progression following 1 to 3 prior lines of anti-neoplastic standard therapy. Therapy in remission after initial induction like intensified chemotherapy for stem cell separation followed by myeloablative therapy or any kind of maintenance therapy is classified as one line of therapy with the induction therapy..
* If Rituximab was part of prior treatment, documented time to progression must be at least 12 weeks after this particular regimen.
* If high-dose Ara-C was part of prior treatment, documented time to progression must be at least 6 months after this particular regimen.
* Patients relapsed after autologous stem cell transplantation or not appropriate for myeloablative treatment.
* At least 1 measurable or assessable site of disease; in case of bone marrow infiltration only, bone marrow aspiration/ biopsy is mandatory for all staging evaluations.
* age > 18 years
* ECOG/WHO Performance Score 0-2 unless lymphoma related.
* The following laboratory values at screening, unless lymphoma related:
* Absolute neutrophil count (ANC) > = 1500 cells/microlitre
* Platelets > = 100,000 cells/microlitre
* Transaminases (AST and ALT) <=3 x upper limit of normal (ULN)
* Total bilirubin <=2 x ULN
* Creatinine <=2 mg/dL or calculated creatinine clearance >=50 mL/min
* Toxic effects of previous therapy or surgery resolved to NCI CTC grade 2 or better.
* Premenopausal fertile females must agree to use a highly effective method of birth control for the duration of the therapy. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
* Men must agree not to father a child for the duration of therapy and must agree to advice a female partner to use a highly effective method of birth control.
* Written informed consent before performance of any study-related procedure.

Exclusion Criteria:

* Previous treatment with Bortezomib
* Treatment within another clinical trial within 30 days before trial entry or planned during this trial
* Anti-neoplastic (including radiation and antibody treatment) or experimental therapy within 4 weeks before planed Day 1 of Cycle 1 (Nitrosoureas within 6 weeks ) or radioimmunoconjugates or toxin immunoconjugates such as Ibritumomab tiuxetan (Zevalin™) or Tositumomab (Bexxar®) within 12 weeks before planed Day 1 of Cycle 1
* Known hypersensitivity to Rituximab, boron or mannitol.
* Active malignancy other than MCL within 5 years before Day 1 of Cycle 1, with the exception of complete resection of basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy.
* Active systemic infection requiring treatment.
* HIV, hepatitis B or C
* Patient has >= grade 2 peripheral sensory neuropathy or neuropathic pain defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE).
* Symptomatic degenerative or toxic encephalopathy
* Serious medical condition (such as severe hepatic impairment, pericardial disease, acute diffuse infiltrative pulmonary disease, systemic infections etc) or psychiatric illness likely to interfere with participation in this clinical study
* Female subject is pregnant or breast-feeding (pregnancy testing is mandatory for premenopausal women).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-05-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline of diseased nodes and nodal masses. | approx. 66 and 126 days after start of therapy
  Average time frame is three weeks after the first two cycles of trial therapy and 4 to 6 weeks after the end of trial therapy.
  Response is always evaluated in comparison to the status before start of trial therapy. The assessment will be done with CT of all known lymphoma manifestations. In case of isolated bone marrow involvement a bone marrow aspiration/ biopsy is mandatory. A minimum of 50 % decrease in SPD (sum of the products of the greatest diameters) of the six largest nodes or nodal masses are necessary, in order to be able to evaluate it as partly remission.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dreyling, MD, Principal Investigator — Klinikum der Universität München, Grosshadern
Locations (54):
- France (21):
  - CH Victor Dupouy, Service hématologie, Argenteuil
  - Centre Hospitalier de la côte Basque, Service hématologie, Bayonne
  - CH de Blois, Service hématologie, Blois
  - Institut Bergonie, Service Hématologie, Bordeaux
  - CH Sud Francilien de Corbeil, Service hématologie, Corbeil-Essonnes
  - Hôpital Henri Mondor, Service hématologie, Créteil
  - Hôpital Albert Michallon, Service hématologie, Grenoble
  - CH Mulhouse, Service hématologie, Le Mans
  - Clinique Victor Hugo, Service hématologie, Le Mans
  - CH du Mans, Service hématologie, Le Mans
  - CHU de Nice, Service hématologie, Nice
  - CHU Necker, Service d'hématologie - adulte, Paris
  - Hôpital Haut Lévêque, Service hématologie, Pessac
  - CHU Lyon Sud, Service hématologie, Pierre-Bénite
  - Hôpital Jean Bernard, Service hématologie, Poitiers
  - CH René Dubos, Service hématologie, Pontoise
  - CHU Robert Debré, Service hématologie, Reims
  - Hôpital Bretonneau, Service hématologie, Bâtiment H. Kaplan, Tours
  - CHU Brabois, Service hématologie, Vandœuvre-lès-Nancy
  - CH de Bretagne Atlantique, Service Hématologie, Vannes
  - Institut Gustave ROUSSY, Villejuif
- Germany (33):
  - Kreisklinik Altötting-Burghausen, Sektion Hämatologie/Onkologie und Palliativmedizin, Altötting
  - Klinikum St. Marien, Med. Klinik II, Amberg
  - Vivantes Klinikum Neukölln, Medizinische Klinik I - Hämatologie und Onkologie, Berlin
  - Knappschaftskrankenhaus, Onkologische Ambulanz, Bottrop
  - Praxis für Hämatologie/Onkologie,, Burgwedel
  - Klinikum der Universität zu Köln, Klinik I f. Innere Medizin, Cologne
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universitätsklinik Essen, Klinik für Hämatologie, Essen
  - Klinikum der J.W. Goethe-Universtität Frankfurt, Medizinische Klinik II, Hämatologie/Onkologie, Frankfurt am Main
  - Ernst-Moritz-Arndt-Universität, Hämatologie/Onkologie, Greifswald
  - Kath. Krankenhaus Hagen gem. GmbH St.-Marien-Hospital, Hagen
  - Asklepios Klinik St. Georg, Abteilung Hämatologie, Hamburg
  - St.-Marien-Hopsital Gem. GmbH, Hamm
  - Universitätsklinik des Saarlandes, Homburg/Saar
  - Westpfalz-Klinikum GmbH, I. Medizinische Klinik, Kaiserslautern
  - UKSH im Städt. Krankenhaus Kiel, II. Med. Klinik und Poliklinik im SSK, Kiel
  - Praxis Dr. Vehling-Kaiser, Landshut
  - Klinikum Magdeburg gemeinnützige GmbH, Klinik f. Hämatologie/Onkologie, Magdeburg
  - Klinikum d. Phillips-Universität, Klinik für Innere Medizin Hämatol./Onkologie/Immunologie, Marburg
  - Kliniken Maria Hilf GmbH (Krankenhaus St. Franziskus), Mönchengladbach
  - Klinikum Schwäbisch Gmünd, Zentrum Innere Medizin, Mutlangen
  - LMU München - Klinikum Großhadern Medizinische Klinik III, München
  - Klinikum Nord Nürnberg, 5. Med. Klinik, Onkologie/Hämatologie, Nuremberg
  - Schlossberg Klinik, Oberstaufen Internistische Onkologie, Oberstaufen
  - Diakonie Klinikum Jung Stilling Krankenhaus, Siegen
  - Diakonieklinikum Stuttgart, Medizinische Klinik II, Stuttgart
  - Robert-Bosch-Krankenhaus, Hämatologie/Onkologie, Stuttgart
  - Mutterhaus der Borromäerinnen, Medizinische Abteilung, Trier
  - Krankenhaus der Barmherzigen Brüder, 1. Medizinische Abteilung, Trier
  - Universitätsklinikum Ulm, Innere Medizin III, Ulm
  - Harz-Klinikum Wernigerode-Blankenburg GmbH, Innere Medizin, Hämato-Onkologie und Palliativmedizin, Wernigerode
  - Ammerland-Klinik GmbH, Klinik für innere Medizin, Westerstede
  - Heinrich-Braun-Krankenhaus, Klinik für Innere Medizin III, Zwickau

REFERENCES:
- [Derived] Fischer L, Jiang L, Durig J, Schmidt C, Stilgenbauer S, Bouabdallah K, Solal-Celigny P, Scholz CW, Feugier P, de Wit M, Trappe RU, Hallek M, Graeven U, Hanel M, Hoffmann M, Delwail V, Macro M, Greiner J, Giagounidis AAN, Dargel B, Durot E, Foussard C, Silkenstedt E, Weigert O, Pott C, Klapper W, Hiddemann W, Unterhalt M, Hoster E, Ribrag V, Dreyling M. The addition of bortezomib to rituximab, high-dose cytarabine and dexamethasone in relapsed or refractory mantle cell lymphoma-a randomized, open-label phase III trial of the European mantle cell lymphoma network. Leukemia. 2024 Jun;38(6):1307-1314. doi: 10.1038/s41375-024-02254-2. Epub 2024 Apr 27. PMID 38678093